CLINICAL TRIAL: NCT07323706
Title: Ayurvedic Diet as a Supplement to Levothyroxine Treatment of Myxedema
Brief Title: Ayurvedic Diet in Myxedema
Acronym: AYUS-MYX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AYUS
Record Dates: First submitted 2025-12-15; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Hypothyroidism Primary
Keywords: hypothyroidism; Vegetarian diet; Ayurveda
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- habitual diet (Other): continuation of habitual diet
  Interventions: Other: habitual diet
- ayurvedic diet (Experimental): plant based ayurvedic diet
  Interventions: Behavioral: Ayurvedic diet

INTERVENTIONS:
Behavioral: Ayurvedic diet — Guidance in implementation of a diet adapted to Vishamagni; which foods and flavors are appropriate to consume, intake of oils, eating patterns, herbal supplements and guidance on which foods and flavors are inappropriate to consume. General Ayurvedic dietary advice for vishamagni: Regular meals; 3 main meals daily at approximately the same time. Consume foods with the Ayurvedic taste nuances: sweet, sour and salty. Primarily consume hot and prepared meals. Eat lactovegetarian. Avoid spicy, bitter and astringent foods. Avoid meat, raw vegetables (all vegetables must be cooked), dry and crunchy foods such as crackers, dried fruit, rice crackers and muesli, and avoid ice cold foods and drinks. One Ayurvedic herbal supplement MA505 (Triphala), with fruits and spices intended to balance the digestive type Vishamagni
  Arms: ayurvedic diet
Other: habitual diet — instruction on continuation of the habitual diet
  Arms: habitual diet

SUMMARY:
Primary hypothyroidism is diagnosed by elevated thyroid stimulating hormone (TSH) level and a reduced thyroxine (T4) level in plasma. Some of the most common symptoms of hypothyroidism are fatigue, weight gain and reduced cognition and is associated with reduced quality of life and increased days of sick leave. Levothyroxine, a synthetic form of T4, is clinically recommended as first-line treatment for hypothyroidism. When normalizing TSH/T4 with levothyroxine, the prevalence of persistent symptoms is present in 15% of patients. The composition of our gut bacteria, the microbiome, plays a significant role for a healthy thyroid gland and metabolism and is influenced by our diet. The Indian medical system, Ayurveda, is based on generations of experience and knowledge in disease prevention and treatment, including various diet plans, exercise and lifestyles that are put into context for physical and mental health. Ayurveda works with four different types of digestion and is based on a vegetarian diet. The purpose of this study is to investigate the effect of an Ayurvedic diet plan, as a supplement to medical treatment, among people with hypothyroidism.

DETAILED DESCRIPTION:
AYURVEDIC DIET AS A SUPPLEMENT TO PHARMACOLOGICAL TREATMENT OF MYXEDEMA

I. INTRODUCTION Hypothyroidism (myxedema) has an estimated prevalence of 3% (1). Mostly women are affected by metabolic diseases in general with a gender distribution of 83% women versus 17% men, according to the Danish Metabolic Association (stofskifteforeningen) (2). Iodine deficiency is a common cause of thyroid diseases, including hypothyroidism. Hashimotos disease (chronic autoimmune thyroiditis) is the primary cause in countries with sufficient iodine (1,3-4), typically requiring lifelong treatment and is partly hereditary affecting across generations (3). Primary hypothyroidism is diagnosed by elevated thyroid-stimulating hormone (TSH) level and a reduced thyroxine (T4) level in plasma (4). Some of the most common symptoms of hypothyroidism are fatigue, cold intolerance and constipation (1,4). Other common symptoms are weight gain, pain in muscles and joints, reduced memory and ability to concentrate, depression as well as hair loss and lack of energy (4). Untreated or undertreated hypothyroidism increases the risk of infertility, neurological and musculoskeletal symptoms, cardiovascular diseases and increased mortality (4-5). Hypothyroidism is associated with reduced quality of life and increased sick leave days (6-11). Levothyroxine, a synthetic form of T4, is clinically recommended as the first-line treatment of hypothyroidism (1,4). The effect target for Levothyroxine treatment is primarily defined based on a normalization of the TSH level (12). This means that the accompanying symptoms can still be present and be a nuisance to the patient, and 15% of patients will continue to have symptoms (7,13), most often reduced cognitive skills and an increased risk of anxiety and depression (14,17) which impair the quality of life (14-18). Even with normalized TSH levels, there is an increased risk of higher BMI and increased use of beta-blockers, statins and antidepressants (19). Most recently, combination treatment with levothyroxine and liothyronine (a synthetic form of T3), as well as treatment with dried thyroid extracts, has attracted great interest, but the effects are still debated, as large randomized clinical studies are lacking and there is uncertainty about the side effect profile (2,20 -21). Recent research has shown that the microbiota affects the metabolism and the thyroid gland (22), and a clear association between the microbiome and our brain function, the so-called gut thyroid axis (23-24) has been shown. Furthermore, it is evident that the composition of the diet is important for the composition of the microbiome (22). For metabolic diseases such as diabetes and overweight, diet planning, so-called medically tailored meals, is used as part of an effective treatment. This also applies to heart disease and chronic liver disease (25). The interest in food as medicine is clear and e.g. the Rockefeller Foundation and the American Heart Association launched a $250 million research initiative (25-27). The microbiome also plays a significant role in a well-functioning thyroid gland and metabolism, and changing the gut bacteria to create dysbiosis increases intestinal permeability. An inflammatory response can thereby occur with proinflammatory cells in the intestines but also in the thyroid (28-29). Dysbiosis is often seen in thyroid patients, where Lactobacillaceae and Bifidobacteriaceae are reduced, which affects the level of thyroid hormones and inhibits TSH (30-31). This may explain the increased comorbidity of thyroid and intestinal diseases (celiac disease and gluten intolerance) (32-35). In addition, the microbiota has an influence on the bioavailability of essential minerals, such as iodine, iron and copper, which are part of the synthesis of thyroid hormones, but also selenium and zinc, which are important for the conversion of T4 to T3. These minerals are often deficient in Hashimoto's thyroiditis, resulting in thyroid malfunction (30,36-38). The Indian medical system, Ayurveda, is based on generations of experience and knowledge in disease prevention and treatment, including various diet plans that are put into context for physical and mental health such as exercise, daily routines and lifestyle (39-42). The interest in Ayurvedic phenotypes (prakriti) has potential for precision medicine, and a study has shown association between these phenotypes and the microbiome (43). It indicates that prakriti (pheno)typing can be a marker for the gut microbiome, which is of importance for an individual's health, disease and treatment (43-44). There are four different Ayurvedic digestive types, agni; Samagni (normal metabolism, agni), Tikshnagni (intense metabolism, agni), Mandagni (mild/weak metabolism, agni) and Vishamagni (irregular metabolism, agni) (40). The digestive types are determined anamnestically based on the digestive pattern; the number of toilet visits per day, the consistency of the stool, appetite, hunger and thirst, acid regurgitation and belching, bloating and flatulence from the intestines as well as pain and pressure in the abdominal area. The most dominant type of digestion, defines the primary type of digestion for an individual, and determines which eating habits, foods and flavors are beneficial and which will be disadvantageous for digestion. The Vishamagni digestive type is considered the easiest to treat, and differs from the other digestive types by being irregular with varying hunger, appetite, thirst, stool pattern, flatulence and belching. In addition, pronounced bloating, pressure and pain in the abdominal area, alternating stools with both hard and loose stools, periodic constipation, exhaustion after meals and varying energy levels are seen (40-41). In comparison, normal digestion is characterized by a balanced appetite, thirst, weight and energy level as well as hunger just before meals and stools 1-2 times a day with normal consistency. In addition, there is no discomfort after meals and no pain, acid regurgitation, flatulence, as well as regular evacuation of air from the intestines and belching (40-41). Ayurveda generally recommends a lacto-vegetarian diet (40-41,45). There is a lack of scientific studies that test the effect of Ayurvedic diet, especially in combination with medical treatment. We wish to generate a pilot study, in order to create scalable effect studies (25).

II. HYPOTHESES A Vishamagni diet plan, as a supplement to medical treatment of hypothyroidism, improves digestion and has a positive effect on frequent symptoms of hypothyroidism, measured by self-reported questionnaire.

III. PURPOSE To investigate the effect of an Ayurvedic Vishamagni diet plan among patients with hypothyroidism. Self-reported changes from before, during and after the treatment are compared for a number of digestion-specific parameters and general health parameters.

IV. METHOD The study is a prospective, exploratory case-control trial in which clients are randomized to follow a Vishamagni or placebo (unchanged) diet plan. The participants are divided, by simple randomization method, into two groups with N participants = 44 in each, where group A receives a Vishamagni diet plan and group B continues the unchanged diet (control group). Both groups A and B must also take a digestion test (oral questions), fill in questionnaires with effect parameters and fill in a diet diary.

Treatment group A One Ayurvedic practitioner, Mette Westerholt, will treat all participants from group A. All participants in group A receive the same treatment and receives 3 consultations in total; 2 treatment consultations and 1 follow-up consultation, which are all held online and 4 weeks apart. The treatment consultations consist of standard Ayurvedic diet recommendations for Vishamagni digestion and one Ayurvedic herbal supplement MA505 (Triphala), with fruits and spices intended to balance the digestive type Vishamagni. No other dietary supplements are taken by the participants.

Treatment consultations 1 and 2: Guidance in implementation of a diet adapted to Vishamagni; which foods and flavors are appropriate to consume, intake of oils, eating patterns, herbal supplements and guidance on which foods and flavors are inappropriate to consume. General Ayurvedic dietary advice for vishamagni: Regular meals; 3 main meals daily at approximately the same time. Consume foods with the Ayurvedic taste nuances: sweet, sour and salty. Primarily consume hot and prepared meals. Eat lactovegetarian. Avoid spicy, bitter and astringent foods. Avoid meat, raw vegetables (all vegetables must be cooked), dry and crunchy foods such as crackers, dried fruit, rice crackers and muesli, and avoid ice cold foods and drinks.

Consultations group B (placebo) One Ayurveda therapist, Mette Westerholt, will carry out all placebo consultations with the participants from group B and consists of 3 conversations without treatment (placebo consultations). The test participants in group B do not consume any kind of nutritional supplements and/or herbs.

V. TRIAL SUBJECTS Inclusion: Women and men of age 18 to 69 who have been diagnosed with primary hypothyroidism, who have primary digestive type Vishamagni, who are under medical treatment for hypothyroidism and who have been stable medicated for the past 6 months.

Exclusion: People with digestive types other than Vishamagni, who have previously been in an Ayurvedic treatment course, who take prescription drugs other than medication for hypothyroidism, as well as pregnant and lactating women.

VII. PROJECT GROUP Mette Westerholt: MSc in Human Biology, University of Copenhagen. 2 years of experience as a scientific assistant on various research projects. Medically examined Ayurvedic health advisor and experience with more than 200 clients in Ayurvedic, individual consultations, including more than 50 clients with hypothyroidism.

Charlotte Bech: International expert and consultant in Ayurvedic diet and lifestyle. Medical doctor with a background in internal medicine. Lecturer at the Danish Parliament and author of 10 books. International expertise through a long-term postgraduate education in India in Maharishi AyurVeda, as well as clinical experience with Maharishi AyurVeda since 2001, in Denmark, Norway and England.

Jens Rikardt Andersen: MD, MPA: Associate Professor in Clinical Nutrition, Department of Sports and Nutrition, University of Copenhagen. Specialist in medical gastrointestinal diseases. Research areas; clinical nutrition, dietary fibers, probiotics, fish oil for the treatment of cancer. Former chairman of the Danish Society for Clinical Nutrition (DSKE).

VIII. LOCATION AND FEASIBILITY The Ayurvedic health consultations take place online, with Mette Westerholt, in the AYUS clinic located in Sorø, Zealand. The study is carried out in a main collaboration between Mette Westerholt at the private company AYUS, collaboration partner doctor Chalotte Bech and main responsible researcher Jens Rikardt Andersen at the Department of Sports and Nutrition, University of Copenhagen. The University of Copenhagen will provide access to all needed software and databases etc.

IX. RESULTS AND PUBLICATION The trial results of the project, positive, negative and inconclusive, are published via www.clinicaltrialsregister.eu. The trial results will be published in peer-reviewed scientific journals.

X. SCIENTIFIC AND SOCIETY-ORIENTED PERSPECTIVES We want to investigate the possibility of alleviating symptoms for patients suffering from hypothyroidism, by implementing dietary changes, and thereby increasing the quality of life, for patients who, despite medication, continue to experience symptoms. In addition, we want to promote the nationwide, western and global acceptance of the Ayurvedic, holistic natural treatment and prevention methods, and create linkage between conventional, evidence-based medicine and the Ayurvedic, holistic health system. We also want to use the identified parameters and effect informatively in future larger and blinded research setups to determine effect size and generalizability.

XI. HOW THE PROJECT ADDRESSES THE APPLIED THEME The main focus of the project is based on patient-related, clinical independent research regarding hypothyroidism that is characterized as a chronic disease that primarily affects women which leads to serious inequality in health between men and women with reduced quality of life for the (mostly female) patient, as well as socio-economic consequences in the form of increased sick leave days. Hypothyroidism can affect all groups of age and typically requires lifelong treatment and is partly hereditary affecting across generations.

REFERENCES

1. Madariaga G.A. et.al. 2014. The incidence and prevalence of thyroid dysfunction in Europe: A meta-analysis. J Clin Endocinol Metab 99(3):923-931.
2. Danish Metabolic Association (Stofskifteforeningen), https://stofskifteforeningen.dk/stofskiftesygdom/lavt-stofskifte/
3. Zaletel K. and Gaberscek S. 2011. Hashimoto's Thyroiditis: From Genes to the Disease. Curr Genomics 12(8):576-588.
4. Chaker L. et.al. 2017. Hypothyroidism. Lancet 390(10101):1550-1562.
5. Thvilum M. et.al. 2013. Excess mortality in patients diagnosed with hypothyroidism: a nationwide cohort study of singletons and twins. J Clin Endocrinol Metabol 98:1069-75.
6. Guglielmi R. et.al. 2018. Shift from levothyroxine tablets to liquid formulation at breakfast improves quality of life of hypothyroid patients. Endocr Metab Immune Disord Drug Targets 18:235-40.
7. Dew R. et.al. 2017. Clinical, behavioural and pharmacogenomic factors influencing the response to levothyroxine therapy in patients with primary hypothyroidism-protocol for a systematic review. Syst Rev 6:60.
8. Ott J. et.al. 2011. Hashimoto´s thyroiditis affects symptom load and quality of life unrelated to hypothyroidism: a prospective case-control study in women undergoing thyroidectomy for benign goiter. Thyroid 21:161-7.
9. Shin Y.W. et.al. 2016. Diminished quality of life and increased brain functional connectivity in patients with hypothyroidism after total thyroidectomy. Thyroid 26:641-9.
10. Vigario P.S. et.al. 2013. Inadequate levothyroxine replacement for primary hypothyroidism is associated with poor health-related quality of life - a Brazilian multicentre study. Endocrine 44:434-40.
11. Thvilum M. et.al. 2014. Hypothyroidism is a predictor of disability pension and loss of labor market income: a danisk register-based study. J. Clin Endocrinol Metabol. 99:3129-35.
12. Laszlo H. et.al. 2022. Primary hypothyroidism and quality of life. Nt Rev Endocrinol. 18(4):230-242.
13. Kraut E. and Farahani P. 2015. A systematic review of clinical practice guidelines recommendations on levothyroxine therapy alone versus combination therapy (LT4 plus LT3) for hypothyroidism. Clin Invest Med. 38:305-13.
14. Wiersinga W.M. et.al. 2012. ETA guidelines: the use of L-T4 + L-T3 in the treatment of hypothyroidism. Eur Thyroid J. 1:55-71.
15. Jonklaas J. et.al. 2014. Guidelines for the treatment of hypothyroidism: prepared by the American thyroid association task force on thyroid hormone replacement. Thyroid 24:1670-1751.
16. Winther K.H. et.al. 2016. Disease-specific as well as generic quality of life is widely impacted in autoimmune hypothyroidism and improes during the first six months of levothyroxine therapy. PloS One 11,e0156925.
17. Saravanan P. et.al. 2002. Psychological well-being in patients on adequate doses of l-thyroxine: results of a large, controlled community-based questionnaire study. Clin. Endocrinol. 57:577-585.
18. Groenewegen K.L. et.al. 2021. Persisting symptoms in patients with Hashimoto´s disease despite normal thyroid hormone levels: Does thyroid autoimmunity play a role? A systematic review. J. Transl. Autoimmun. 4,100101.
19. Peterson S.J. 2016. Is a normal TSH synonymous with "euthyroidism" in levothyroxine monotherapy? J Clin Endocrinol Metab 101:4964-4973.
20. Jonklaas J. et.al. 2021. Evidence-based use of levothyroxine/liothyronine combinations in treating hypothyroidism: a consensus document. Eur. Thyroid J. 10:10-38.
21. La Cour J.L. et.al. 2022. Socioeconomic influences treatment with liothyronine and desiccated thyroid extract in Denmark. Eur Thyroid J. 11(6):e220149.
22. Hills R.D. et.al. 2019. Gut microbiome: Profound implications for diet and disease. Nutrients 11(7):1613.
23. Bargiel P. et.al. 2021. Microbiome metabolites and thyroid dysfunction. J Clin Med 10(16):3609.
24. Jiang W. et.al. 2022. The relationship between the gut microbiota and its metabolites with thyroid diseases. Front Endocrinol 13: 943408.
25. No authers listed. 2023. Food as medicine: translating the evidence. Nature Medicine 29(4):753-754.
26. Teong X.T. et.al. 2023. Intermittent fasting plus early time-restricted eating versus calorie restriction and standard care in adults at risk of type 2 diabetes: a randomized controlled trial. Nature Medicine 29:963-962.
27. Watanabe K. et.al. 2023. Multiomic signatures of body mass index identify heterogeneous health phenotypes and responses to a lifestyle intervention. Nature Medicine 29(4):1-13.
28. Frölich, E. and Wahl R. 2019. Microbiota and thyroid interaction in health and disease. Trends Endocrinol. Metab. 30:479-490.
29. Lerner A. et.al. 2017. Gut-thyroid axis and celiac disease. Endocr. Connect. 6:52-58.
30. Knezevic J. et.al. 2020. Thyroid-Gut-Axis: How does the microbiota influence thyroid function. Nutrients 12(6):1769
31. Nguyen T.T. et.al. 1993. 5´- and 5-deiodinase activities in adult rat cecum and large bowel contents inhibited by intestinal microflora. Am. J. Physiol. Metab. 265:521-524.
32. Kahaly G.J. et.al. 2018. Celiac disease and glandular autoimmunity. Nutrients 10:814.
33. Roy A. et.al. 2016. Prevalence of celiac disease in patients with auatoimmune thyroid disease: A meta-analysis. Thyroid 26: 880-890.
34. Losurdo G. et.al. 2015. Evolution of nonspecific duodenal lymphocytosis over 2 years of follow-up. World J. Gastroenterol. 21:7545-7552.
35. Volta U. et.al. 2014. An Italian prospective multicenter survey on patients suspected of having non-celiac gluten sensitivity. BMC Med. 12:85.
36. Zimmermann M.B. and Boelaert K. 2015. Iodine deficiency and thyroid disorders. Lancet Diabetes Endocrinol 3(4):286-95.
37. Wozniak D. et.al. 2021. Dietary supplements in hypothyroidism. Acta Sci Pol Technol Aliment 20(4):375-381.
38. Zhou Q. et.al. 2022. Trace elements and the thyroid. Front Endocrinol 24:13:904889.
39. Gokani T. 2014. Ayurveda - the science of healing. Headache 54(6):1103-6.
40. R.K. Sharma and B. Dash (Eds. and Trans.): Caraka Samhita (Caraka Samhita Vol. 1,2,3,4,5,6 and 7). Chowkhamba Press, Varanasi, India: Chowkhamba Sanskrit Series (1988), Vol. XCIV.
41. Sebastian Pole. 2013. Ayurvedic Medicine, The Principles of Traditional Practice. Churchill Livingstone, Elsevier.
42. Patwardhan B. 2014. Bridging Ayurveda with evidence-based scientific approaches in medicine. EPMA 5(1):19.
43. Chauhan Nar S. et.al. 2018. Western Indian Rural Gut Microbial Diversity in Exteme Prakriti Endo-Phenotypes Reveals Signature Microbes. Frontiers in Microbiology 9(118):1-12.
44. Jnana A. et.al. 2020. Prakriti phenotypes as a stratifier of gut microbiome: A new frontier in personalized medicine? Journal of Ayurveda and Integrative Medicine 11:360-365.
45. Wallac R.K. 2020. The Microbiome in Health and Disease from the Perspective of Moderne Medicine and Ayurveda. Medicina (Kaunas) 11;56(9):462.
46. Singh A. et.al. 2017. Development, validation, and verification of a self-assessment tool to estimate Agnibala (digestive strength). Journal of evidence-based complementary & alternative medicine 22(1):134-140.
47. Edwards M.T. and Streiner D.L. 2022. Development of a reliable dosha self-assessment questionnaire. Explore 18(5):573-578.
48. Eswaran H.T. et.al. 2015. Formation and validation of questionnaire to assess Jätharäghi. Ancient Science of Life 34(4):203-209.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with primary hypothyroidism
* primary digestive type Vishamagni
* under medical treatment for hypothyroidism
* unchanged medication for the past 6 months

Exclusion Criteria:

* previous Ayurvedic treatment
* prescription drugs other than medication for hypothyroidism
* pregnancy
* lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
digestion | 8 weeks
  change in digestion measured by self-reported questionnaire

SECONDARY OUTCOMES:
symptoms of hypothyroidis | 8 weeks
  symptoms of hypothyroidism measured by self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, MPA, Study Chair — University of Copenhagen; Mette Westerholt, MSc, Principal Investigator — AYUS
Locations (2):
- Denmark (2):
  - Department of Nutrition, Exercise and Sports, Copenhagen, Frederiksberg
  - Ayuvedic Clinic, Sorø, Sorø

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://ayus.dk/ayurvedisk-forskningsprojekt/